CLINICAL TRIAL: NCT01881308
Title: REmission in Rheumatoid Arthritis - Assessing WIthrawal of Disease-modifying Antirheumatic Drugs in a Non-inferiority Design
Brief Title: Assessing Withdrawal of Disease-Modifying Antirheumatic Drugs in Rheumatoid Arthritis
Acronym: ARCTIC REWIND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Research Council of Norway (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Espen A. Haavardsholm, MD PhD, MD PhD, Head of Department, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIA2012-1/ver4_1; 2012-005275-14 (EudraCT Number)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Stable dose TNF inhibitor (Active Comparator): Stable dose TNF inhibitor. Any co-medication with synthetic DMARDs kept stable.
  Interventions: Drug: TNF inhibitors; Drug: Co-medication: Synthetic DMARDs
- Stepdown and withdrawal of TNF inhibitor (Experimental): Half-dose of TNF inhibitor for the first four months, thereafter withdrawal of TNF inhibitor. Any co-medication with synthetic DMARDs kept stable.
  Interventions: Drug: TNF inhibitors; Drug: Co-medication: Synthetic DMARDs
- Stable dose synthetic DMARD (Active Comparator): Stable dose of synthetic DMARDs, either monotherapy or combination therapy.
  Interventions: Drug: Synthetic DMARD(s)
- Synthetic DMARD dose reduction (Experimental): Half-dose synthetic DMARDs (monotherapy or combination therapy) for the first 12 months of the study. Patients classified as non-failures are re-randomized at 12 months to either continue half-dose synthetic DMARD(s) or withdraw all DMARD(s).
  Interventions: Drug: Synthetic DMARD(s)
- ARCTIC follow-up (Other): Patients are treated according to the ARCTIC treatment schedule based on disease activity.
  Interventions: Drug: TNF inhibitors; Drug: Synthetic DMARD(s); Drug: Co-medication: Synthetic DMARDs

INTERVENTIONS:
Drug: TNF inhibitors
  Arms: ARCTIC follow-up; Stable dose TNF inhibitor; Stepdown and withdrawal of TNF inhibitor
Drug: Synthetic DMARD(s)
  Arms: ARCTIC follow-up; Stable dose synthetic DMARD; Synthetic DMARD dose reduction
Drug: Co-medication: Synthetic DMARDs — Synthetic DMARDs given as co-medication for TNF inhibitors as appropriate.
  Arms: ARCTIC follow-up; Stable dose TNF inhibitor; Stepdown and withdrawal of TNF inhibitor

SUMMARY:
The purpose of this study is to assess the effect of disease-modifying anti-rheumatic drugs (DMARDs) dose reduction in patients with rheumatoid arthritis (RA).

Remission is the treatment target in RA, but knowledge about the best way to treat RA patients who achieve sustained remission is limited. DMARDs have potential serious adverse events, and biologic DMARDs are costly to the society. The objectives for ARCTIC REWIND are to assess the effect of tapering and withdrawal of DMARDs on disease activity in RA patients in sustained remission, to study predictors for successful tapering and withdrawal of DMARDs in this patient group, and to study cost-effectiveness of different treatment options in RA remission.

ARCTIC REWIND is a randomized, open, controlled, parallel-group, multicenter, phase IV, non-inferiority strategy study. Patients with less than five years of disease duration and stable remission for at least 12 months are randomized to either continued stable treatment or tapering and withdrawal of DMARDs, including tumor necrosis factor (TNF) inhibitors and synthetic DMARDs. Patients are assessed by clinical examination, patient reported outcome measures, ultrasonography, MRI and X-ray, and monitored for adverse events. The primary endpoint of the study is the proportion of patients who are non-failures (have not experienced a flare) at 12 months. Secondary endpoints include composite disease activity scores and remission criteria, joint damage and inflammation assessed by various imaging modalities, work participation, health care resource use and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria
* Male or non-pregnant, non-nursing female
* >18 years of age and <80 years of age
* Patient in the TNF-inhibitor group: Any disease duration. Patient in the synthetic DMARD group: RA diagnosis after 01.01.2010.
* Sustained remission for ≥12 months according to DAS or Disease Activity Score based on 28 joints (DAS28), with documented remission status at a minimum of 2 consecutive visits during the last 18 months OR participation in the first ARCTIC trial
* DAS <1.6 and no swollen joints at inclusion OR participation in the first ARCTIC trial
* Unchanged treatment with TNF inhibitors and/or synthetic DMARDs during the previous 12 months, with a stable or reduced dose of glucocorticosteroids OR participation in the first ARCTIC trial
* Subject capable of understanding and signing an informed consent form
* Provision of written informed consent

Exclusion Criteria:

* Abnormal renal function, defined as serum creatinine >142 μmol/L in female and >168 μmol/L in male, or a glomerular filtration rate (GFR) <40 mL/min/1.73 m2
* Abnormal liver function (defined as aspartate transaminase (ASAT)/alanine aminotransferase (ALAT) >3x upper normal limit), active or recent hepatitis, cirrhosis
* Major co-morbidities, such as severe malignancies, severe diabetic mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class 3 or 4) and/or severe respiratory diseases
* Leukopenia and/or thrombocytopenia
* Inadequate birth control, pregnancy, and/or breastfeeding
* Indications of active tuberculosis
* Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol impossible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are non-failures (have not experienced a flare) | 12 months
  Flare is defined as composite measure: (1) An increase in disease activity score (DAS) to >1.6 AND (2) a change in DAS of at least 0.6 AND (3) > 1 swollen joint. If a patient does not fulfill this formal definition, but experiences a clinically significant flare according to the investigator and patient, this is treated as a flare.

SECONDARY OUTCOMES:
Disease Activity Score (DAS) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The DAS is a composite score that includes the Ritchie articular index (RAI), the 44- swollen joint counts (SJC-44), the Erythrocyte Sedimentation Rate (ESR) and a general health (GH) assessment on a Visual Analogue Scale (VAS).
  The DAS is calculated as follows:
  DAS = 0.54*sqrt(RAI) + 0.065*(SJC-44) + 0.33*Ln(ESR) + 0.0072*GH
Disease Activity Score in 28 joints (DAS28) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The 28-joint Disease Activity Score (DAS28) includes the 28- tender joint counts (TJC28), 28-swollen joint counts (SJC28), Erythrocyte Sedimentation Rate (ESR) and Patient Global Assessment (PGA) on a VAS.
Simplified Disease Activity Index (SDAI) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  SDAI includes TCJ28, SJC28, PGA, physician's global assessment of disease activity on a VAS 0-100 mm (PhGA) and C-reactive protein (CRP).
Clinical Disease Activity Index (CDAI) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  CDAI includes TCJ28, SJC28, PGA and PhGA.
Swollen joint count | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Swollen joint counts are performed on 44 joints, with total joint count ranging from 0 to 44.
Tender joint count | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Tender joints is assessed by Ritchie Articular Index which assesses tenderness of 26 joint regions, based on summation of joint responses after applying firm digital pressure. The index ranges from 0 to 3 for individual measures and the sum 0 to 78 overall.
Erythrocyte Sedimentation Rate (ESR) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Assessment of ESR in mm/h
C-reactive protein (CRP) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Assessment of CRP in mg/L
Patient's assessment of disease activity (PGA) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  PGA is the patient's assessment of disease activity on a VAS 0-100 mm.
Physician's global assessment of disease avtivity (PHGA) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  PHGA is the investigator's assessment of disease activity on a VAS 0-100 mm.
Health Assessment Questionnaire (HAQ-PROMIS) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The HAQ-PROMIS is a questionnaire evaluating the physical function in patients with RA.
EuroQol-5 Dimension (EQ-5D) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.
Medical Outcomes Study Short-Form 36-item (SF-36) Physical and Mental Component Summary Score | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Work performance | 12 months, with subsequent long-term analyses after 24 months and 36 months
  1. Absenteeism (work time missed)
  2. Presenteeism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivity loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment
Radiographic joint damage | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Radiographs of hands (posterior/anterior) and foot (anterior/posterior) will be taken at baseline, 12, 24 and 36 months. The modified Sharp van der Heijde Score (vdHSS) will be calculated, including an erosion score and a joint space narrowing score.
Ultrasonography (subclinical synovitis) | 12 months, with subsequent long-term analyses after 24 months and 36 months
  36 joints and 2 tendons will be scored for both grey scale and power doppler synovitis on a 0-3 scale.
DAS-remission | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Remission is defined as a DAS-score <1.6
DAS28-remission | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Remission is defined as a DAS28 score < 2.6
SDAI-remission | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Remission is defined as a SDAI score ≤ 3.3
CDAI-remission | 12 months, with subsequent long-term analyses after 24 months and 36 months
  Remission is defined as a CDAI score ≤ 2.8
ACR/EULAR Boolean remission | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The patient must satisfy all of the following in order to achieve ACR/EULAR remission:
  * RAI ≤ 1
  * SJC44 ≤ 1
  * CRP ≤ 1
  * PGA ≤ 1 (on a scale 0-10, in this study ≤ 14 on a scale 0-100)
No swollen joint | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The percentage of patients with no swollen joints will be assessed
Radiographic outcome | 12 months, with subsequent long-term analyses after 24 months and 36 months
  No radiographic progression
Ultrasound outcome | 12 months, with subsequent long-term analyses after 24 months and 36 months
  No ultrasound power Doppler signal in any joint.
American College of Rheumatology (ACR) response | 12 months, with subsequent long-term analyses after 24 months and 36 months
  If a patient has experienced a flare, and treatment has been escalated, the ACR 2050/70/90 response will be calculated.
The European League Against Rheumatism (EULAR) response | 12 months, with subsequent long-term analyses after 24 months and 36 months
  If a patient has experienced a flare, and treatment has been escalated, the EULAR response will be calculated.
The Food and Drug Administration (FDA) major clinical response | 12 months, with subsequent long-term analyses after 24 months and 36 months
  If a patient has experienced a flare, and treatment has been escalated, the FDA major clinical response will be calculated.
Medication | 12 months, with subsequent long-term analyses after 24 months and 36 months
  The number of patients on different conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) and biologic therapy. Dose of DMARDs in users will be recorded, prednisolone usages and number of intraarticular injections.

CONTACTS AND LOCATIONS:
Overall Officials: Espen A. Haavardsholm, MD PhD, Principal Investigator — Diakonhjemmet Hospital; Tore K Kvien, MD PhD, Study Director — Diakonhjemmet Hospital
Locations (10):
- Norway (10):
  - Department of Rheumatology, Helse Møre og Romsdal HF, Ålesund
  - Department of Rheumatology, Haukeland University Hospital, Helse Bergen HF, Bergen
  - Department of Rheumatology, Drammen Hospital, Vestre Viken HF, Drammen
  - Department of Rheumatology, Sykehuset Østfold HF, Fredrikstad
  - Department of Rheumatology, Sørlandet Sykehus HF, Kristiansand
  - Revmatismesykehuset AS, Lillehammer
  - Helgelandssykehuset, Mo i Rana, Mo i Rana
  - Department of Rheumatology, Diakonhjemmet Hospital, Oslo
  - Martina Hansens Hospital AS, Sandvika
  - Universitetssykehuset Nord-Norge HF, Tromsø

IPD SHARING:
Plan to Share IPD: Yes
The authors commit to making the relevant anonymized patient level data available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by the study steering committee, and requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Kjorholt KE, Sundlisaeter NP, Aga AB, Sexton J, Olsen IC, Fremstad H, Spada C, Madland TM, Hoili CA, Bakland G, Lexberg A, Hansen IJW, Hansen IM, Haukeland H, Ljosa MA, Moholt E, Uhlig T, Kvien TK, Solomon DH, van der Heijde D, Haavardsholm EA, Lillegraven S. Effects of tapering conventional synthetic disease-modifying antirheumatic drugs to drug-free remission versus stable treatment in rheumatoid arthritis (ARCTIC REWIND): 3-year results from an open-label, randomised controlled, non-inferiority trial. Lancet Rheumatol. 2024 May;6(5):e268-e278. doi: 10.1016/S2665-9913(24)00021-3. Epub 2024 Apr 4. PMID 38583450
- [Derived] Holten K, Paulshus Sundlisaeter N, Sexton J, Nordberg LB, Uhlig T, Kvien TK, Solomon DH, Haavardsholm EA, Lillegraven S, Aga AB; ARCTIC REWIND study group. Performance of the Rheumatoid Arthritis Impact of Disease (RAID) score in relation to flares in disease activity. RMD Open. 2024 Jan 12;10(1):e003486. doi: 10.1136/rmdopen-2023-003486. PMID 38216290
- [Derived] Lillegraven S, Paulshus Sundlisaeter N, Aga AB, Sexton J, Olsen IC, Lexberg AS, Madland TM, Fremstad H, Hoili CA, Bakland G, Spada C, Haukeland H, Hansen IM, Moholt E, Uhlig T, Solomon DH, van der Heijde D, Kvien TK, Haavardsholm EA. Effect of tapered versus stable treatment with tumour necrosis factor inhibitors on disease flares in patients with rheumatoid arthritis in remission: a randomised, open label, non-inferiority trial. Ann Rheum Dis. 2023 Nov;82(11):1394-1403. doi: 10.1136/ard-2023-224476. Epub 2023 Aug 22. PMID 37607809
- [Derived] Lillegraven S, Paulshus Sundlisaeter N, Aga AB, Sexton J, Olsen IC, Fremstad H, Spada C, Madland TM, Hoili CA, Bakland G, Lexberg A, Hansen IJW, Hansen IM, Haukeland H, Ljosa MA, Moholt E, Uhlig T, Solomon DH, van der Heijde D, Kvien TK, Haavardsholm EA. Effect of Half-Dose vs Stable-Dose Conventional Synthetic Disease-Modifying Antirheumatic Drugs on Disease Flares in Patients With Rheumatoid Arthritis in Remission: The ARCTIC REWIND Randomized Clinical Trial. JAMA. 2021 May 4;325(17):1755-1764. doi: 10.1001/jama.2021.4542. PMID 33944875